CLINICAL TRIAL: NCT02989961
Title: Autologous Intra-lesional Injection of Resticutis Compared to Platelet-Poor Plasma to Improve Healing of Wagner's Grade II/III Diabetic Foot Ulcers (Neuropathic/Neuro-Iscemic)
Brief Title: Safety and Efficacy of Resticutis Compared to Platelet-Poor Plasma for Treating Diabetic Foot Ulcers
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hanan Jafar (Other)
Responsible Party: Sponsor-Investigator, Hanan Jafar, Researcher, University of Jordan
Organization: University of Jordan (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Resticutis.UJCTC
Record Dates: First submitted 2016-11-29; First posted 2016-12-12 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A-Resticutis (Experimental): Autologous, Activated-Platelets type of preparation.
  Interventions: Other: Resticutis
- C-Platelet-Poor Plasma PPP (Placebo Comparator): Platelet-Poor Plasma type of preparation achieved by centrifugation of blood samples at high speed conditions. Resticutis is administered instead if the patient doesn't achieve full healing after 6 injections.
  Interventions: Other: Resticutis; Other: Platelet-Poor Plasma (PPP)

INTERVENTIONS:
Other: Resticutis — Autologous, Activated-Platelets type of Preparation
  Other Names: Actiplate 1
Other: Platelet-Poor Plasma (PPP) — A preparation of low platelet plasma obtained by a high-speed centrifugation step.
  Arms: C-Platelet-Poor Plasma PPP

SUMMARY:
The purpose of this study is to determine the safety of Resticutis for the treatment of Wagner's Grade II/III diabetic foot ulcers in comparison with Platelet-Poor Plasma as a placebo comparator.

DETAILED DESCRIPTION:
Grade II and III (According to Wagner's classification system of Ulcer severity) are considered to be of the most common complications associated with Diabetes, which are mostly hard to heal using the conventional treatment methods which by consequence severely affects the quality and lifestyle of the diabetes patient.

It's thought that the application of Autologous activated platelets "Resticutis" which secretes huge amounts of growth factors is capable of giving better results of which are: the stimulation of the healing process that includes contraction, granulation, tissue formation and epithelialization of the diabetic foot ulcer.

Resticutis is obtained from an autologous 20 mL peripheral blood withdrawn in tubes containing 3.8% Sodium Citrate. Blood is then centrifuged to obtain Platelet-Rich Plasma -PRP- as per established method. PRP is then activated in a closed system by physical methods to obtain a final product of 5 mL of Resticutis which is injected intra-lesionally at ulcer margins per each session of therapy.

It's hypothesized that a total of six injections throughout the period of the treatment are enough to achieve full closure of the DFU. The injections are given on days: 0,14,28,42,56, and 70 of the treatment period.

The consenting patients will be randomized into 2 groups: One group will be given Resticutis, and the second one Platelet-Poor Plasma PPP as placebo. If patients in PPP group didn't achieve full healing after four-six injections, they're given a two weeks rest after which they are given Resticutis instead.

This is mainly a phase 1 safety study, which means no formal statistical analysis will be applied to any of the data. Safety assessment will depend on the association of any adverse events during the course of the study, and efficacy as a secondary objective will be assessed by observing the healing time of DFUs.

ELIGIBILITY:
Inclusion Criteria:

* People with Type II Diabetes mellitus between the ages of 18 and 70 with an ulcer with at least 4 weeks duration.
* Hb1c of less than 13 %.
* Index foot ulcer located on the plantar, medial, or lateral aspect of the foot (including all toe surfaces), and wound area (length*width) measurement between 0.5 cm^2 and 20 cm^2, inclusive.
* Wounds located under a Charcot deformity has to be free of acute changes and went through appropriate structural consolidation.
* Wagner Grade II or III ulcer.
* The protocol requires that post-debridement, the ulcer would be free of necrotic debris, foreign bodies, or sinus tracts.
* Non invasive vascular testing Ankle Brachial Index (ABI).
* Physical examination (Including a Semmes-Weinstein monofilament test for neuropathy).
* Blood tests to be obtained (CBC, Hb1c)
* Approved, informed, signed consent to be obtained from each patient.

Exclusion Criteria:

* Patient currently enrolled in another investigative device or drug trial or previously enrolled (within the last 30 days) in an investigative research of a device or a pharmaceutical agent.
* Ulcer area decreased > 50% during the seven-day screening period.
* Ulcer is due to a non-diabetic etiology.
* Evidence of gangrene in ulcer or on any part of the foot.
* Patient is currently receiving or has received radiation or chemotherapy within the last 3 months of randomization.
* Patient has received growth factor therapy within 7 days of randomization.
* Screening platelets count < 100* 10^9/L.
* Patient is undergoing renal dialysis, or has a known immune insufficiency, known abnormal platelets activation disorder (i.e. Grey Platelet Syndrome, Liver Disease, Active Cancer), eating/nutritional, hematologic, collagen vascular disease, rheumatic disease, or bleeding disorder.
* History of peripheral vascular repair within 30 days of randomization.
* Patient is known to have a physiological, developmental, physical, emotional, or social disorder, or any other situation that may interfere with their compliance with the study requirements and/or the healing of the ulcer.
* History of alcohol or drug abuse within the last year prior to randomization.
* Patient has inadequate venous access for blood withdraw.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-11-15 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) as a result of the injection | 2 months
  Evaluate the safety of this treatment, by gathering and assessing the number, timing, severity, duration, and resolution of related adverse events.

SECONDARY OUTCOMES:
Assess the efficacy of autologous Resticutis injection by clinical examination | 4 months
  To determine short term speed and effectiveness of autologous Resticutis as a platelet lysate derivative on the healing of diabetic foot ulceration compared with Platelet Poor Plasma by measuring the healing time.

IPD SHARING:
Plan to Share IPD: No